CLINICAL TRIAL: NCT05849649
Title: Increasing Physical Activity Through a Mobile Health Intervention Among Pregnant and Postpartum Women in a Rural Setting
Brief Title: Mobile Application-based Exercise Intervention for Pregnant Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western Kentucky University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB 20-257
Record Dates: First submitted 2023-03-29; First posted 2023-05-09 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-11

CONDITIONS: Pregnancy Related; Postpartum
Keywords: exercise; mHealth; pregnancy; postpartum; rural
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BumptUp Mobile App (Experimental): The intervention group will have full access to the BumptUp mobile app which includes exercise and dietary progress tracking, social support, evidence-based and safe exercise programming, videos, and symptom tracking.
  Interventions: Behavioral: BumptUp
- Educational Brochure/ Attention Control (Active Comparator): This group will receive evidence-based exercise education the form a one-time brochure.
  Interventions: Behavioral: Educational Brochure

INTERVENTIONS:
Behavioral: BumptUp — The app contains a number of evidence-based, expertly designed features to help women with healthier lifestyle habits during and after pregnancy.
  Arms: BumptUp Mobile App
Behavioral: Educational Brochure — An evidence-based brochure on physical activity
  Arms: Educational Brochure/ Attention Control

SUMMARY:
The overarching goal of this randomized controlled clinical trial is to test the efficacy of the mHealth app (BumptUp) for improving physical activity levels among pregnant and postpartum women in a rural setting. Secondary outcomes include weight status, dietary intake, glucose tolerance, blood pressure, and mental health.

Specific Aim 1. Conduct an RCT (N=176) to assess the efficacy of the mHealth intervention for increasing physical activity levels during pregnancy (13-15, 23-25, and 35-37 weeks gestation) and postpartum (6 and 12 weeks) among women in a rural setting.

Research Activities: The efficacy of BumptUp® will be determined by measuring physical activity levels (via accelerometry and surveys) between women who use the mobile app (intervention) and women who use only an educational brochure (attention control).

Specific Aim 2: Assess the efficacy of the mHealth intervention on important obstetric outcomes including maternal weight status, dietary intake, glucose tolerance, blood pressure, and mental health.

Research Activities: Maternal weight status, glucose tolerance, and blood pressure values will be obtained from patient charts. Dietary intake will be assessed via the National Cancer Institute Multifactor Screener. Maternal mental health status will be measured via The Edinberg Postpartum Depression Questionnaire, Center for Epidemiological Studies Depression Scale, and the State-Trait Anxiety Inventory.

DETAILED DESCRIPTION:
A mobile application (app) that can increase physical activity during and after pregnancy is novel, timely, and critically important to maternal health. Mobile phone-based interventions show significant promise because they can be tailored to the target population, can be delivered at any place and at any time (with or without internet connection), are interactive, and are accessible to the majority of the population irrespective of socioeconomic status (96% of U.S. women ages 18-49 own smartphones). The use of mHealth apps has been associated with behavior change, specifically adaptation of healthy lifestyle approaches. The majority of pregnant women report using an app related to pregnancy; it is the health condition with the highest number of apps available. However, high-quality evidence-based mobile apps that address physical activity specifically for pregnancy do not exist. The overarching goal of this randomized controlled clinical trial is to test the efficacy of the mHealth app for improving physical activity levels among pregnant and postpartum women in a rural setting. Secondary outcomes include weight status, dietary intake, glucose tolerance, blood pressure, and mental health.

After contact is established and eligibility confirmed, participants (N=176) will undergo a screener, a baseline assessment, and then randomized to the mHealth intervention or the attention control group. All participants will have data collected at the following timepoints: baseline (13-15 weeks pregnant), mid-pregnancy (23-25 weeks), late pregnancy (35-37 weeks), and postpartum (6 and 12 weeks). [Of note, 12-week interventions during pregnancy are customary and have been shown to elicit clinically meaningful changes in outcomes. The pilot study protocol was 12 weeks of pregnancy and 12 weeks postpartum.] The proposed RCT will add an additional timepoint in early pregnancy (13-15 weeks), which will increase the length of the intervention to 39+ weeks. This will further enhance the likelihood of the intervention influencing behavior and outcomes.

There will also be three check-ins via telephone (two during pregnancy and one during postpartum upon medical clearance at ~6 weeks) to aid with retention, as well as allow participants to ask any questions about the app (intervention) or the educational brochure (attention control). The 13-15 week gestation time point was chosen because most women have had an initial prenatal appointment (to ensure viability) and the risk of miscarriage substantially reduced. The late pregnancy timepoint was selected as women tend to become the least active during late pregnancy. Six weeks postpartum was selected as this is when most women have their only postpartum clinical appointment (i.e. opportunity for objective clinical data extraction). The 12-week time point is important for assessing behavior as women transition back into activity after medical clearance, which is important for long-term sustained activity.

After the baseline assessment (13-15 weeks gestation), the women will be randomized to the intervention or attention control group. The intervention group will receive free access to the mobile app (BumptUp®). BumptUp® users will watch an introductory video on the app's features which reiterates the goal of the app: to reach the recommended 150 minutes per week of physical activity. The app contains evidence-based workout information and education as well as several resources aimed at increasing physical activity and overcoming barriers for women during and after pregnancy. Each app feature is not only developed as the result of feedback from rural study participants, but is developed with a specific mechanism for behavior change in mind.

The attention control group will undergo the exact same study protocol (parallel) and receive the same amount of interaction from the study team; however, participants will obtain an electronic evidence-based educational brochure about physical activity and dietary intake during pregnancy instead of access to BumptUp®. To ensure the control group is a true attention control, the study team has paid careful attention to recommendations and will ensure that the control group receives the exact same amount of interpersonal interaction as intervention participants (same number of emails, phone calls, surveys, and face-to-face interactions). Instead of a tutorial on the app at the time of randomization, participants will have an educational session with the study team about the educational brochure.

Data Collected at each timepoint: To assess the primary outcome of physical activity (Aim 1), participants will wear an Actigraph wGT3X-BT Accelerometer (ActiGraph LLC,) on their wrist for seven consecutive days at each time point (Pregnancy: 13-15 weeks, 23-25 weeks, 35-37 weeks, Postpartum: 6 and 12 weeks). Monitoring physical activity for one week at multiple time points is standard in exercise research. Actigraph provides an accurate and reliable way to assess overall physical activity levels. Wrist-worn tri-axel accelerometers are a valid measure of physical activity in pregnant women. Data will be collected for seven consecutive days at 30Hz. The accelerometer output will be sampled by a 12-bit analog-to-digital converter. Categories of activity will be determined using the following cut points: Sedentary (0-99counts/minute), light (100-1951 counts/min), moderate (1952-5724 counts/minute), and vigorous (≥5725 counts/min). The percentage of time spent sedentary as well as the amount of time spent participating in different categories of physical activity ranging from light to vigorous will be calculated. Non-wear times will be excluded from the analyses. Women will be asked to wear the devices for seven consecutive days without removal. If removed, it must be documented it so the study team can be sure it does not interfere with the analyses. The study team has a successful history of compliance with these devices among pregnant women, including the pilot study for the present intervention. Devices will be dropped off with careful instructions for when/how to wear the device and when/how to remove it. Because many women in the study reside in rural areas, the accelerometer can be delivered by mail with a prepaid return envelope to increase compliance. Because all participants will receive prenatal care at one of two clinics, prenatal appointments will also be utilized to meet participants and deliver/pick up accelerometer devices. Physical activity will also be assessed subjectively using the Exercise Vital Sign survey-a survey specifically designed to determine whether someone meets 150 minutes of physical activity per week (i.e. meets the recommendations from the ACOG).

The same participants and study design will be followed for Aim 2. The outcomes of focus for this aim will be obstetric outcomes with clear links to maternal morbidity and mortality rates, including maternal weight status, glucose tolerance, blood pressure, and mental health.

Medical data will be collected directly from patient charts in order to assess will be used to determine weight status, glucose tolerance, and blood pressure. Team members (Dr. Maire Blankenship and Dr. Leigh Lindsey) will pull data directly from the Graves Gilbert Clinic and Women's Health Specialist's electronic medical record systems. These data include height, weight, and blood pressure results at prenatal appointments that correspond to data collection time points (i.e., 12-17 weeks, 23-27 weeks (wider time ranges due to appointments still being monthly for many women during early-to-mid pregnancy), 35-37 weeks, and 6-weeks postpartum. All data at 12 weeks postpartum will be patient/participant self-report as there are no routine postpartum visits at 12 weeks. Per standard-of-care clinical protocols, oral glucose tolerance testing occurs at 24-28 weeks gestation and will be used to determine glucose tolerance. Extracted data will be used to determine the impact of the intervention on weight gain/retention, blood pressure, and glucose tolerance. The study team has already been granted permission to collect these data (see letters of support) and has a history of success at collecting these assessments per the pilot project.

To assess mental health, electronic surveys will be distributed at each time point. These include the Edinberg Postpartum Depression Questionnaire and the State-Trait Anxiety Inventory. Maternal depression and anxiety play a significant role in maternal morbidity and mortality, and physical activity improves symptoms of both during and after pregnancy. Therefore, it is important to understand if the mHealth app improves mental health. Research clearly shows a need to assess both anxiety and depression during and after pregnancy, as anxiety tends to be more common and more often overlooked. Therefore, the State-Trait Anxiety Inventory was chosen to measure anxiety. Further, it is exceedingly clear that exercise can assist with reducing anxiety. In order to assess the app's ability to improve dietary intakes, as well as account the possible confounding impact of dietary intake on weight status, the National Cancer Institute Multifactor (Diet) Screener will be provided as part of the electronic survey package.

At each time point, surveys will be administered via Research Electronic Data Capture (REDCap). During the pilot, data were successfully collected, and exit interviews indicate an acceptable level of participant burden.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-44
* Confirmed singleton viable pregnancy
* English-Speaking (the app is currently only available in English)
* Physician release to participate in exercise prior to study participation
* Ownership of a smartphone
* Patient at either Graves Gilbert Clinic or Women's Health Specialists
* Plans to deliver at The Medical Center in Bowling Green, KY.

Exclusion Criteria:

* Multiple gestation pregnancy
* Inability to provide voluntary informed consent
* Any medical condition (pregnancy-related or not) that would preclude exercise.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 176 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Physical activity level (objective) | 13-15 weeks gestation
  Measured via Actigraph accelerators
Physical activity level (objective) | 23-25 weeks gestation
  Measured via Actigraph accelerometer
Physical activity level (objective) | 35-37 weeks gestation
  Measured via Actigraph accelerometer
Physical activity level (subjective) | 6 weeks postpartum
  Measured via Exercise Vital Signs (survey)
Physical activity level (objective) | 12 weeks postpartum
  Measured via Actigraph accelerometer
Physical activity level (subjective) | 13-15 weeks gestation
  Exercise Vital Sign Survey
Physical activity level (subjective) | 23-25 weeks gestation
  Exercise Vital Sign Survey
Physical activity level (subjective) | 35-37 weeks gestation
  Exercise Vital Sign Survey
Physical activity level (subjective) | 12 weeks postpartum
  Exercise Vital Sign Survey

SECONDARY OUTCOMES:
Maternal Weight Status | 13-15 weeks gestation
  Measured via objective medical chart data on maternal weight
Maternal Weight Status | 23- 25 weeks gestation
  Measured via objective medical chart data on maternal weight
Maternal Weight Status | 35-37 weeks gestation
  Measured via objective medical chart data on maternal weight
Maternal Weight Status | 6 weeks postpartum
  Measured via objective medical chart data on maternal weight
Maternal Weight Status | 12 weeks postpartum
  Self-reported weight data
Dietary Intake | 13-15 weeks gestation
  The National Cancer Institute Multifactor Screener
Dietary Intake | 23-25 weeks gestation
  The National Cancer Institute Multifactor Screener
Dietary Intake | 35-37 weeks gestation
  The National Cancer Institute Multifactor Screener
Dietary Intake | 6 weeks postpartum
  The National Cancer Institute Multifactor Screener
Dietary Intake | 12 weeks postpartum
  The National Cancer Institute Multifactor Screener
Glucose Tolerance | 24-28 weeks gestation
  Oral Glucose Tolerance test results obtained from routine clinical assessments and extracted from charts
Blood Pressure (systolic and diastolic) | 13-15 weeks gestation
  Extracted from clinical charts
Blood Pressure (systolic and diastolic) | 23-25 weeks gestation
  Extracted from clinical charts
Blood Pressure (systolic and diastolic) | 35-37 weeks gestation
  Extracted from clinical charts
Blood Pressure (systolic and diastolic) | 6 weeks postpartum
  Extracted from clinical charts
Mental Health (Depression) | 13-15 weeks gestation
  The Edinberg Postpartum Depression Questionnaire (Minimum value:0, maximum value 30). Higher scores indicate a worse outcome/more likely to be depressed. Anything over 12 is considered to have depression.
Mental Health (Depression) | 23-35 weeks gestation
  The Edinberg Postpartum Depression Questionnaire (Minimum value:0, maximum value 30). Higher scores indicate a worse outcome/more likely to be depressed. Anything over 12 is considered to have depression.
Mental Health (Depression) | 35-37 weeks gestation
  The Edinberg Postpartum Depression Questionnaire (Minimum value:0, maximum value 30). Higher scores indicate a worse outcome/more likely to be depressed. Anything over 12 is considered to have depression.
Mental Health (Depression) | 6 weeks postpartum
  The Edinberg Postpartum Depression Questionnaire (Minimum value:0, maximum value 30). Higher scores indicate a worse outcome/more likely to be depressed. Anything over 12 is considered to have depression.
Mental Health (Depression) | 12 weeks postpartum
  The Edinberg Postpartum Depression Questionnaire (Minimum value:0, maximum value 30). Higher scores indicate a worse outcome/more likely to be depressed. Anything over 12 is considered to have depression.
Mental Health (Anxiety) | 13-15 weeks gestation
  State-Trait Anxiety Inventory
Mental Health (Anxiety) | 23-25 weeks gestation
  State-Trait Anxiety Inventory. This is a 40-question survey using a 4-point Likert Scale ranging from almost never to almost always. Scores for both State Anxiety and Trait Anxiety (20 questions each) range from 20 to 80, with higher scores indicating higher levels of anxiety.
Mental Health (Anxiety) | 35-37 weeks gestation
  State-Trait Anxiety Inventory This is a 40-question survey using a 4-point Likert Scale ranging from almost never to almost always. Scores for both State Anxiety and Trait Anxiety (20 questions each) range from 20 to 80, with higher scores indicating higher levels of anxiety.
Mental Health (Anxiety) | 6 weeks postpartum
  State-Trait Anxiety Inventory This is a 40-question survey using a 4-point Likert Scale ranging from almost never to almost always. Scores for both State Anxiety and Trait Anxiety (20 questions each) range from 20 to 80, with higher scores indicating higher levels of anxiety.
Mental Health (Anxiety) | 12 weeks postpartum
  State-Trait Anxiety Inventory This is a 40-question survey using a 4-point Likert Scale ranging from almost never to almost always. Scores for both State Anxiety and Trait Anxiety (20 questions each) range from 20 to 80, with higher scores indicating higher levels of anxiety.
Neonatal Body Composition | 24-48 hours post-delivery
  Air Displacement Plethysmography (Bod Pod)
Neonatal body fat percentage | 24-48 hours post-delivery
  Skinfold Calipers (4 site method)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel A Tinius, PhD, Principal Investigator — Western Kentucky University
Locations (1):
- Rachel Tinius, Bowling Green, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No